CLINICAL TRIAL: NCT06298084
Title: Phase 1b/2, Multicenter, Open-label, Dose-Expansion Modular Study To Explore the Safety, Tolerability, and Anti-tumor Activity of HER3- DXd Monotherapy and Combinations in Patients With Inoperable Advanced Breast Cancer (ABC) After Progression on T-DXd
Brief Title: Dose-Expansion Modular Study To Explore the Safety, Tolerability, and Anti-tumor Activity of HER3- DXd Monotherapy and Combinations in Patients With Inoperable Advanced Breast Cancer (ABC) After Progression on T-DXd
Acronym: ICARUSBREAST02
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2023-505925-15-00; 2023/3668 (Other: CSET number)
Record Dates: First submitted 2024-02-12; First posted 2024-03-07 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer Metastatic; HER2-positive Metastatic Breast Cancer; HER2 Low Breast Carcinoma; Advanced Breast Cancer
MeSH Terms: interventions — patritumab deruxtecan; olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part 1a (safety run-in module 0) (Experimental): Patients with HER2-low ABC who have progressed on T-DXd. Patients in part 1a will receive intravenous infusion of HER3-DXd monotherapy (5.6 mg/kg every 21 days)
  Interventions: Drug: Patritumab deruxtecan
- Part 1b (dose finding module 1 + dose expansion module 0) (Experimental): In the dose expansion part, patients will receive the RP2D defined in the dose finding part of different combinations (module 1) and HER3-DXd single agent 5.6 mg/kg IV D1 every 21 days in module 0.
  Interventions: Drug: Patritumab deruxtecan; Drug: Olaparib
- Part 2 (dose expansion module 1 + module 0) (Experimental): In the dose expansion part, patients will receive the RP2D defined in the dose finding part of different combinations (module 1) and HER3-DXd single agent 5.6 mg/kg IV D1 every 21 days in module 0.
  Interventions: Drug: Patritumab deruxtecan; Drug: Olaparib

INTERVENTIONS:
Drug: Patritumab deruxtecan — 5.6 mg/kg every 21 days
  Other Names: U3-1402; HER3-DXd
Drug: Olaparib — 100 mg b.i.d PO days 8-14 every 21 days
  Other Names: Lynparza
  Arms: Part 1b (dose finding module 1 + dose expansion module 0); Part 2 (dose expansion module 1 + module 0)

SUMMARY:
ICARUS-BREAST02 is an open-label, multicenter, phase 1b/2, platform study that aims to evaluate the safety, tolerability, and efficacy of HER3-DXd monotherapy and in combination with other anti-cancer agents in patients with ABC.

The first 2 modules will evaluate: i. safety and efficacy of HER3-DXd with olaparib in patients with HER2-low and HER2-positive ABC progressed on T-DXd (Module 1) and HER3-DXd monotherapy in patients with HER2-low ABC progressed on T-DXd (Module 0).

The main objective of Part 1 is to assess the safety and tolerability of HER3-DXd monotherapy and combination and to determine the recommended phase 2 dose (RP2D) of the combination containing HER3-DXd.

The main objective of Part 2 is to assess the efficacy of study therapies in each module based on investigator assessment as evaluated by the objective response rate (ORR) at 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have received prior treatment with T-DXd and presented disease progression while on T-DXd treatment or within 2 months from T-DXd interruption/discontinuation for any reason, without requiring to be the last line of treatment. Patients who have received other lines of treatment after T-DXd and before study entry is capped at 10 patients for each cohort.
2. Patients with HER2-positive tumors must have received prior treatment with trastuzumab and taxanes. They may have received prior treatment with T-DM1 and pertuzumab.
3. Patients with HER2-low tumors must have been treated with taxanes. Patients with HR-positive tumors must have received ET and CDK4/6 inhibitors (patients may have received prior treatment with sacituzumab govitecan) If a patient has a tumor that was previously HER2-pos and became HER2-low, she/he will be included in cohort 2 and meet the inclusion criteria for HER2-low tumors.

   If a patient has a tumor that was previously HR-pos and became HR-neg, prior therapy with CDK4/6 inhibitors is not mandatory.
4. Patients with germline pathogenic BRCA1/2 mutations and HER2-positive or HER2-low breast cancer are eligible to the study but must have received a prior treatment with PARP inhibitor (olaparib or talazoparib)
5. Female or male patient aged ≥18 years on the day of the ICF signature
6. Patient who has histologically confirmed diagnosis of breast cancer with unresectable loco regional or metastatic disease
7. Patient must have an ECOG PS ≤1 at the time of screening
8. Patients must have HER2-pos (IHC 3+ or IHC2+/ISH positive) or HER-2 low (IHC2+/ISH negative or IHC 1+) tumors with any HR status, any time before T-DXd exposure
9. Patient must have at least one radiologically measurable lesion (different from the biopsy site) according to response evaluation criteria in solid tumors (RECIST) V1.1 criteria. At least one predominantly lytic or mixed lytic-blastic bone lesion with identifiable soft tissue component that can be evaluated by Computerized Tomography (CT)/Magnetic Resonance Imaging (MRI) must be present in patients with only bone metastasis
10. Patient must have a tumor site easily accessible to biopsy, avoiding bone biopsy when possible. Patients must have accepted to perform pre-treatment, on-treatment, and end-of-treatment biopsies
11. Patient must have adequate bone marrow reserve and organ function, based on local laboratory data within 14 days prior to Cycle 1, Day 1, defined per the protocol
12. Female patients of reproductive/childbearing potential must have a negative pregnancy test at screening (serum test within 24 hours before C1D1 or urine test within 72 hours of C1D1) and must and must agree to use a highly effective form of contraception or avoid intercourse during and till the end of treatment and for at least 8 months after the last dose of study drug. The following contraception methods are considered highly effective:

    1. Intrauterine device (IUD)
    2. Bilateral tubal occlusion
    3. Vasectomized partner
    4. Complete sexual abstinence defined as refraining from heterosexual intercourse during and till the end of treatment and for at least 8 months for females after the last dose of study drug. Periodic abstinence not an acceptable method of contraception
13. Female patients must not donate, or retrieve for their own use, ova from the time of screening and throughout the study treatment period, and for at least 8 months after the final study drug administration
14. Male patients must be surgically sterile or must withhold heterosexual intercourse, or must be willing to use a highly effective birth control upon enrollment, during the treatment period, and for at least 5 months following the last dose of study drug
15. Male patients must not freeze or donate sperm starting at screening and throughout the study period, and for at least 5 months after the final study drug administration.
16. Patient must understand, sign and date the written informed consent form (ICF) prior to any protocol-specific procedures performed. Patient should be able and willing to comply with study visits and procedure as per protocol
17. Patient must be affiliated to a social security system or beneficiary of the same

Exclusion Criteria:

The following exclusion criteria are applicable for all modules. Patients will be excluded if they present one of them:

1. Patient with a breast cancer amenable for resection or radiation therapy with curative intent
2. Patient with any history of ILD (including pulmonary fibrosis or radiation pneumonitis), has current ILD, or is suspected to have ILD as assessed by imaging during screening
3. Patient with clinically severe pulmonary compromise (based on investigator's assessment) resulting from intercurrent pulmonary illnesses including, but not limited to:

   1. Any underlying pulmonary disorder (eg, pulmonary embolism, severe asthma, severe chronic obstructive pulmonary disease (COPD), restrictive lung disease, pleural effusion) OR
   2. Any autoimmune, connective tissue or inflammatory disorder with pulmonary involvement (eg, rheumatoid arthritis, Sjögren's syndrome, sarcoidosis) OR
   3. Prior pneumonectomy
4. Patient receiving chronic systemic corticosteroids dosed at >10 mg/day prednisone or equivalent anti-inflammatory activity or any form of immunosuppressive therapy prior to Cycle 1 Day 1. Patients who require use of bronchodilators, inhaled or topical steroids, or local steroid injections may be included in the study
5. Patient with evidence of any leptomeningeal disease
6. Patient with clinically significant corneal disease
7. Patient with any evidence of severe or uncontrolled systemic diseases (e.g. active bleeding diatheses, active infection, or psychiatric illness) which in the investigator's opinion makes it undesirable for the patient to participate in the study or which would jeopardize compliance with the protocol. Screening for chronic conditions is not required for eligibility
8. Evidence of spinal cord compression or brain metastases, defined as being clinically active and symptomatic, or requiring therapy with corticosteroids or anticonvulsants to control associated symptoms. Patients with clinically inactive or treated brain metastases who are asymptomatic (ie, without neurologic signs or symptoms and do not require treatment with corticosteroids or anticonvulsants) may be included in the study. Patients must have a stable neurologic status for at least 2 weeks prior to Cycle 1 Day 1
9. Inadequate washout period prior to Cycle 1 Day 1, defined as:

   1. Whole brain radiation therapy or stereotactic brain radiation therapy <14 days
   2. Previous treatment with T-DXd < 28 days
   3. Any cytotoxic chemotherapy, investigational agents or other anticancer drug(s) from a previous cancer treatment regimen or clinical study <14 days or 5 half-lives, whichever is longer
   4. Endocrine therapy <21 days
   5. Monoclonal antibodies <28 days including immune checkpoint inhibitors (ICIs)
   6. Major surgery (excluding placement of vascular access) <28 days
   7. Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation <28 days or palliative radiation therapy <14 days
   8. Live virus vaccination <28 days
10. Prior treatment with an anti-HER3 antibody
11. Patients with unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet resolved to grade ≤1 or baseline, as defined by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. Patients with chronic Grade 2 toxicities (defined as no worsening to Grade >2 for at least 3 months prior to enrollment and managed with standard of care treatment) that the Investigator deems related to previous anticancer therapy, comprising the following, may be enrolled at the discretion of the Investigator:

    * Chemotherapy-induced neuropathy
    * Fatigue
    * Residual toxicities from prior immuno-oncology treatment: Grade 1 or Grade 2 endocrinopathies provided they are clinically stable and receiving hormone replacement therapy when applicable which may include:

      1. Hypothyroidism/ hyperthyroidism
      2. Type I diabetes
      3. Hyperglycemia
      4. Adrenal insufficient
      5. Adrenalitis
      6. Skin hypopigmentation (vitiligo)
12. Has known hypersensitivity to either the drug substances or the inactive ingredients of HER3-DXd and/or T-DXd
13. Patient with a history of severe hypersensitivity reactions to other monoclonal antibodies or PARP inhibitors
14. Has any malignancy other than locally advanced or ABC within 3 years prior to Cycle 1 Day 1, except adequately resected non-melanoma skin cancer or curatively treated in-situ disease or other curatively treated solid tumors
15. Documented uncontrolled or significant cardiovascular disorder prior to Cycle 1 Day 1, including:

    1. Corrected QT interval >450 ms according to Fridericia's formula (QTcF) based on triplicate 12-lead ECGs, approximately 1 minute apart
    2. LVEF <45% by either ECHO or MUGA or cardiac MRI if clinically indicated according to the investigator or consulting cardiologist
    3. Resting systolic blood pressure >140 mmHg or diastolic blood pressure >90 mmHg
    4. Myocardial infarction within 6 months
    5. Symptomatic congestive heart failure (NYHA class from III to IV)
    6. Uncontrolled angina pectoris within 6 months
    7. Cardiac arrhythmia not controlled by ongoing antiarrhythmic treatment
    8. Diagnosed or suspected long QT syndrome, or known family history of long QT syndrome
    9. History of clinically relevant ventricular arrhythmias, such as ventricular tachycardia, ventricular fibrillation, or Torsade de Pointes
    10. Patient has bradycardia of less than 50 bpm (as determined by central reading) unless the subject has a pacemaker
    11. History of second or third degree heart block. Candidates with a history of heart block may be eligible if they currently have pacemakers, and have no history of fainting or clinically relevant arrhythmia with pacemakers
    12. Coronary/peripheral artery bypass graft within 6 months
    13. Complete left bundle branch block
16. Active Hepatitis B and/or Hepatitis C infection, such as those with serologic evidence of active viral infection within 28 days of Cycle 1, Day 1. Patients with past or resolved Hepatitis B virus (HBV) infection are eligible if:

    1. Hepatitis B surface antigen (HBsAg) negative and hepatitis B core antibody (anti-HBc) positive; OR
    2. HBsAg positive and HBV deoxyribonucleic acid (DNA) viral load is documented to be ≤ 2000 IU/mL in the absence of anti-viral therapy and during the previous 12 weeks prior to the viral load evaluation with normal transaminases (in the absence of liver metastasis); OR
    3. HBsAg positive and HBV DNA viral load is documented to be ≤2000 IU/mL in the absence of anti-viral therapy and during the previous 12 weeks prior to the viral load evaluation with liver metastasis and abnormal transaminases AST/ALT <3 ULN For patients with HBsAg positive, if abnormal liver function is detected during study drug treatment, viral load should be tested to rule out reactivation.

    Patients with a history of Hepatitis C infection will be eligible for enrollment only if the viral load according to local standards of detection, is documented to be below the level of detection in the absence of anti-viral therapy during the previous 12 weeks (ie, sustained viral response according to the local product label but not less than 12 weeks, whichever is longer)
17. Female patient who is pregnant or breastfeeding or intends to become pregnant during the study
18. Has a known human immunodeficiency virus (HIV) infection that is not well controlled. All the following criteria are required to define an HIV infection that is well controlled: undetectable viral ribonucleic acid (RNA) load, CD4+ counts/levels of >350 cells/μL, no history of acquired immunodeficiency syndrome (AIDS)-defining opportunistic infection within the past 12 months, and stable for at least 3 weeks on same anti-HIV retroviral medications. If an HIV infection meets the above criteria, the patient's viral RNA load and CD4+ cell count should be monitored per local standard of care (eg, every 3 months). Patients with a well-controlled HIV infection may only be enrolled into Part 2 (dose expansion) of the study.
19. Prior or ongoing clinically relevant illness, medical condition, surgical history, physical finding, or laboratory abnormality that, in the Investigator's judgment, could affect the safety of the patient; alter the absorption, distribution, metabolism or excretion of the study drug; or confound the assessment of study results
20. Adult under legal protection: guardianship, curatorship, or legal protection; or patient deprived of his/her liberty by a judicial or administrative decision; or patient incapable of giving his/her consent, or patient under psychiatric care
21. Participation in another clinical trial evaluating an experimental drug during the last 4 weeks (except non-interventional research) Specific exclusion criteria for each module

    Module 0:

    There are no specific exclusion criteria for module 0 (HER3-DXd monotherapy). Module 1 (olaparib)
22. History of hypersensitivity to excipients of olaparib
23. Inadequate washout period prior to Cycle 1 Day 1, defined as:

    1. Strong CYP3A inhibitors < 1 week
    2. CYP3A inducers for olaparib and phenobarbital < 5 weeks and for any other drug < 3 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2024-03-21 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
DLTs (dose-limiting toxicity) for part 1a and 1b | 21 months after the beginning of enrolment
  DLTs
Frequency of safety event for part 1a and 1b | 21 months after the beginning of enrolment
  frequency of any AEs, TEAEs, SAEs, AESIs graded by NCI-CTCAE v5.0
Severity of safety event for part 1a and 1b | 21 months after the beginning of enrolment
  severity of any AEs, TEAEs, SAEs, AESIs graded by NCI-CTCAE v5.0
Proportion of treatment modification due to AEs for part 1a and 1b | 21 months after the beginning of enrolment
  Proportion of treatment discontinuations, interruptions, and dose reductions due to any AEs
frequency of laboratory abnormalities for part 1a and 1b | 21 months after the beginning of enrolment
  frequency of laboratory abnormalities defined by NCI-CTCAE v5.0 laboratory findings
Severity of laboratory abnormalities for part 1a and 1b | 21 months after the beginning of enrolment
  Severity of laboratory abnormalities defined by NCI-CTCAE v5.0 laboratory findings
radiographic changes potentially consistent with ILD/pneumonitis or any other pulmonary signs/symptoms for part 1a and 1b | 21 months after the beginning of enrolment
  Evaluations must include CT (preferably high-resolution CT) and pulmonologist consultation (when the Investigator is not a pulmonologist). Those will be reviewed by an internal multidisciplinary team at GRCC.
ORR for part 2 | 51 months
  ORR is defined as the proportion of patients who achieved a confirmed complete response (CR) or partial response (PR) assessed by investigators after 6 months of treatment initiation. The objective response will be radiologically assessed every 6 weeks during the first year than every 12 weeks thereafter using RECIST v1.1.
DOR for part 2 | 51 months
  DOR is defined as the time from the date of the first documentation of confirmed response (CR or PR) to the date of the first documentation of progression (PD) or death due to any cause, whichever occurs first. Duration of response will be measured for responding patients (CR or PR) only
PFS for part 2 | 51 months
  PFS is defined as the time from date of first dose until the date of the first objective documentation of disease progression or death from any cause, whichever occurs first. For patients without documented radiological progression, PFS will be censored at the date of last adequate radiological assessment without progression
CBR for part 2 | 51 months
  CBR is defined as the presence of at least a confirmed PR or CR, or a stable disease (SD) ≥ 6 months

SECONDARY OUTCOMES:
ORR for part 1 | 45 months
  ORR is defined as the proportion of patients who achieved a confirmed complete response (CR) or partial response (PR) assessed by investigators after 6 months of treatment initiation. The objective response will be radiologically assessed every 6 weeks during the first year than every 12 weeks thereafter using RECIST v1.1.
DOR for part 1 | 45 months
  DOR is defined as the time from the date of the first documentation of confirmed response (CR or PR) to the date of the first documentation of progression (PD) or death due to any cause, whichever occurs first.Duration of response will be measured for responding patients (CR or PR) only
PFS for part 1 | 45 months
  PFS is defined as the time from date of first dose until the date of the first objective documentation of disease progression or death from any cause, whichever occurs first. For patients without documented radiological progression, PFS will be censored at the date of last adequate radiological assessment without progression.
CBR for part 1 | 45 months
  CBR is defined as the presence of at least a confirmed PR or CR, or a stable disease (SD) ≥6 months
PK analysis for part 1 | 45 months
  Serum concentration of HER3-DXd (Anti-HER3-ac-DXd total, anti-HER3 antibody and DXd), plasma concentration of olaparib, will be assessed for PK analysis. Estimation of the proportion of deconjugated payload-linker complex binding with circulating albumin will also be assessed.
ADA analysis for part 1 | 45 months
  Serum concentration of HER3-DXd (Anti-HER3-ac-DXd total, anti-HER3 antibody and DXd), plasma concentration of olaparib, will be assessed for incidence and prevalence of anti-drug antibody (ADA) for HER3-DXd. Estimation of the proportion of deconjugated payload-linker complex binding with circulating albumin will also be assessed.
DLTs for part 2 | 39 months from the beginning of enrolment
Frequency of safety event for part 2 | 39 months from the beginning of enrolment
  Frequency of any AEs, TEAEs, SAEs, AESIs graded by NCI-CTCAE v5.0;
Severity of safety event for part 2 | 39 months from the beginning of enrolment
  Frequency of any AEs, TEAEs, SAEs, AESIs graded by NCI-CTCAE v5.0;
proportion of treatment modification event for part 2 | 39 months from the beginning of enrolment
  proportion of treatment discontinuations, interruptions, and dose reductions due to any AEs
frequency of laboratory abnormalities for part 2 | 39 months from the beginning of enrolment
  frequency of laboratory abnormalities defined by NCI-CTCAE v5.0;
Severity of laboratory abnormalities for part 2 | 39 months from the beginning of enrolment
  Severity of laboratory abnormalities defined by NCI-CTCAE v5.0;
radiographic changes potentially consistent with ILD/pneumonitis or any other pulmonary signs/symptoms for part 2 | 39 months from the beginning of enrolment
  Evaluations must include CT (preferably high-resolution CT) and pulmonologist consultation (when the Investigator is not a pulmonologist). Those will be reviewed by an internal multidisciplinary team at GRCC.
PK analysis for part 2 | 39 months from the beginning of enrolment
  Serum concentration of HER3-DXd (Anti-HER3-ac-DXd total, anti-HER3 antibody and DXd), plasma concentration of olaparib, will be assessed for PK analysis. Estimation of the proportion of deconjugated payload-linker complex binding with circulating albumin will also be assessed.
ADA analysis for part 2 | 39 months from the beginning of enrolment
  Serum concentration of HER3-DXd (Anti-HER3-ac-DXd total, anti-HER3 antibody and DXd), plasma concentration of olaparib, will be assessed incidence and prevalence of anti-drug antibody (ADA) for HER3-DXd. Estimation of the proportion of deconjugated payload-linker complex binding with circulating albumin will also be assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy Institut, Villejuif, France